CLINICAL TRIAL: NCT05967923
Title: Effectiveness of Shock Wave Therapy Versus Low Level Lazer Therapy in Diabetic
Brief Title: Effectiveness of Shock Wave Therapy Versus Low Level Lazer Therapy in Diabetic Frozen Shoulder Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T- ORTH-06/2023-516
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Complications
Keywords: Diabetes; Frozen shoulder
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Bursitis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Group (a) Group (b) Group (c)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (a) (Experimental): Patients in this group will receive shock wave therapy once a week for four weeks in addition to routine physical therapy program.
  Interventions: Radiation: Shock wave therapy; Other: Routine physical therapy program
- Group (b) (Experimental): Patients in this group will receive low level lazer therapy three times per week for four weeks in addition to routine physical therapy program.
  Interventions: Radiation: Low level lazer therapy; Other: Routine physical therapy program
- Group (c) (Experimental): Patients in this group will receive only routine physical therapy program.
  Interventions: Other: Routine physical therapy program

INTERVENTIONS:
Radiation: Shock wave therapy — Patients in this group will receive shock wave therapy once a week for four weeks in addition to routine physical therapy program.
  Other Names: Non
  Arms: Group (a)
Radiation: Low level lazer therapy — Patients in this group will receive low level lazer therapy three times a week week for four weeks in addition to routine physical therapy program.
  Other Names: Non
  Arms: Group (b)
Other: Routine physical therapy program — Patients in this group will receive only routine physical therapy program three times a week for four weeks.

SUMMARY:
Patients will be divided randomly into 3 groups.

DETAILED DESCRIPTION:
Patients will be allocated from out patient clinics of Qena university hospitals Then they will be randomly assigned to three groups, every one will contain 30 patients of both gender, with age range between 45 and 60 years old

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes mellitus.
* patients with frozen shoulder due to diabetes mellitus.
* patients age ranged between 45 and 60 years old.
* cooperative patients.

Exclusion Criteria:

* patients with un-controlled hypertension.
* patients sensetive to shock wave or lazer irradiation.
* Patients with infectious skin diseases.
* un-cooperative patients.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder joint Pain | 4 weeks
  By using visual analogue scale
Range of motion of the shoulder | 4 weeks
  Range of shoulder internal and external rotation and shoulder flexion

SECONDARY OUTCOMES:
Shoulder and hand disability | 4 weeks
  By using quick DASH questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shymaa yussuf abo zaid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No